CLINICAL TRIAL: NCT04645693
Title: The Impact of Oral Health on Metabolism and Persistent Inflammation in HIV Patients on Antiretroviral Therapy
Brief Title: The Impact of Oral Health in HIV Patients on Antiretroviral Therapy
Acronym: OHART
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Temitope Omolehinwa, BDS, DScD, Assistant Professor of Oral Medicine, University of Pennsylvania
Other Study IDs: 843328; R01DE029648-01 (NIH)
Record Dates: First submitted 2020-10-01; First posted 2020-11-27 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: HIV; Periodontal Diseases; Caries; Non-communicable Disease; Xerostomia
MeSH Terms: conditions — Periodontal Diseases; Noncommunicable Diseases; Xerostomia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — saliva, oral swab and blood samples will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV Subjects with Non-Communicable Diseases: Patients living with HIV on Antiretroviral Therapy drugs for at least one year with no diagnosis of non-communicable diseases (diabetes, insulin resistance, hyperlipidemia/dyslipidemia, vascular disease, and/or osteoporosis).
- HIV Subjects without Non-Communicable Diseases: Patients living with HIV on Antiretroviral Therapy drugs for at least one year with a diagnosis of one or more systemic non-communicable diseases (diabetes, insulin resistance, hyperlipidemia/dyslipidemia, vascular disease, and/or osteoporosis).

SUMMARY:
This is a prospective cohort study designed to investigate the range of metabolic abnormalities observed in patients living with HIV on antiretroviral therapy. This study will also explore the concurrent role of poor oral health in supporting and driving chronic immune activation and inflammation in HIV infection.

DETAILED DESCRIPTION:
This is a prospective cohort study designed to investigate the range of metabolic abnormalities observed in patients living with HIV (PLWH) on antiretroviral therapy (ART). This study will also explore the concurrent role of poor oral health in supporting and driving chronic immune activation and inflammation in HIV infection.

Following enrollment in study, patients will be followed up every 6 months for approximately 2.5 years (30 months). During this period, comprehensive medical records will be obtained, and study data will be updated every 6 months; questionnaires will be handed to patients periodically to assess quality of life and effects of xerostomia on QoL; social history will be assessed using TAPS; oral health will be evaluated every 6 months and blood, saliva, and oral swabs collected every 6 months. DXA scan and panoramic radiographs will also be taken at baseline and 24 months.

At the end of the study, caries rate, periodontal health, bone loss, QoL, salivary quantity and composition, presence or absence of white/red lesions, as well as inflammatory cytokines and immune activation markers will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Has been diagnosed with HIV (as documented by a prior laboratory report of positive HIV-1/2 antibody and/or detectable HIV RNA, available for review by the study team)
* Has received antiretroviral therapy for at least 12 months
* Able and willing to provide informed consent prior to initiation of study procedures
* Willing and able to comply with all study procedures, and likely to be available for the duration of the study

Exclusion Criteria:

* Has been diagnosed with the following xerostomia-related autoimmune conditions: Sjorgen's and sarcoidosis
* Has never received radiation therapy to the head or neck (including radioactive iodine therapy)
* Was taking anti-osteoporotic agents (biphosphonates, denosumab) prior to HIV diagnosis.
* Women who are pregnant at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living with HIV above the age of 18 will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dental Caries as assessed by DMFS Score | Baseline
  Decayed, missing and filled surfaces (DMFS) score to assess dental caries. Minimum value is 0 and maximum value is 128 for 28 teeth. Higher scores mean higher levels of dental decay.
Dental Caries as assessed by DMFS Score | 6 months after baseline visit
  Decayed, missing and filled surfaces (DMFS) score to assess dental caries. Minimum value is 0 and maximum value is 128 for 28 teeth. Higher scores mean higher levels of dental decay.
Dental Caries as assessed by DMFS Score | 12 months after baseline visit
  Decayed, missing and filled surfaces (DMFS) score to assess dental caries. Minimum value is 0 and maximum value is 128 for 28 teeth. Higher scores mean higher levels of dental decay.
Dental Caries as assessed by DMFS Score | 18 months after baseline visit
  Decayed, missing and filled surfaces (DMFS) score to assess dental caries. Minimum value is 0 and maximum value is 128 for 28 teeth. Higher scores mean higher levels of dental decay.
Dental Caries as assessed by DMFS Score | 24 months after baseline visit
  Decayed, missing and filled surfaces (DMFS) score to assess dental caries. Minimum value is 0 and maximum value is 128 for 28 teeth. Higher scores mean higher levels of dental decay.
Dental Caries as assessed by DMFS Score | 30 months after baseline visit
  Decayed, missing and filled surfaces (DMFS) score to assess dental caries. Minimum value is 0 and maximum value is 128 for 28 teeth. Higher scores mean higher levels of dental decay.
Periodontal disease | Baseline
  Incidence of periodontal disease
Periodontal disease | 12 months after baseline visit
  Incidence of periodontal disease
Periodontal disease | 24 months after baseline visit
  Incidence of periodontal disease
Periodontal disease | 30 months after baseline visit
  Incidence of periodontal disease
Oral mucosal lesions coinfection as assessed by the presence or absence of candidiasis, red/white lesions, ulcers and warts intraorally | Baseline
  Prescence or absence of warts, red or white lesions and candidia
Oral mucosal lesions coinfection as assessed by the presence or absence of candidiasis, red/white lesions, ulcers and warts intraorally | 6 months after baseline visit
  Prescence or absence of warts, red or white lesions and candidia
Oral mucosal lesions coinfection as assessed by the presence or absence of candidiasis, red/white lesions, ulcers and warts intraorally | 12 months after baseline visit
  Prescence or absence of warts, red or white lesions and candidia
Oral mucosal lesions coinfection as assessed by the presence or absence of candidiasis, red/white lesions, ulcers and warts intraorally | 18 months after baseline visit
  Prescence or absence of warts, red or white lesions and candidia
Oral mucosal lesions coinfection as assessed by the presence or absence of candidiasis, red/white lesions, ulcers and warts intraorally | 24 months after baseline visit
  Prescence or absence of warts, red or white lesions and candidia
Oral mucosal lesions coinfection as assessed by the presence or absence of candidiasis, red/white lesions, ulcers and warts intraorally | 30 months after baseline visit
  Prescence or absence of warts, red or white lesions and candidia
Osteopenia as assessed by DXA scan findings | Baseline
  Incidence of osteopenia
Osteopenia as assessed by DXA scan findings | 24 months after baseline visit
  Incidence of osteopenia
Quality of life as assessed by the Xerostomia Quality of Life Scale (XeQoLS) | Baseline
  The XeQoLS consists of 15 questions. The first 14 questions assess how dryness in the mouth impacts the individual's life, with answer options of "not at all," "a little," "somewhat," "quite a bit," and "very much." The final question asks "if you were to spend the rest of your life with your dry mouth/throat dryness just the way it is now, how would you feel about this?" and includes options ranging from "delighted" to "terrible." All 15 questions can be translated to a score of 0-4, with a score of 4 indicating the most dry mouth-related problems and 0 indicating no dry mouth-related problems.
Quality of life as assessed by the Xerostomia Quality of Life Scale (XeQoLS) | 12 months after baseline visit
  The XeQoLS consists of 15 questions. The first 14 questions assess how dryness in the mouth impacts the individual's life, with answer options of "not at all," "a little," "somewhat," "quite a bit," and "very much." The final question asks "if you were to spend the rest of your life with your dry mouth/throat dryness just the way it is now, how would you feel about this?" and includes options ranging from "delighted" to "terrible." All 15 questions can be translated to a score of 0-4, with a score of 4 indicating the most dry mouth-related problems and 0 indicating no dry mouth-related problems.
Quality of life as assessed by the Xerostomia Quality of Life Scale (XeQoLS) | 24 months after baseline visit
  The XeQoLS consists of 15 questions. The first 14 questions assess how dryness in the mouth impacts the individual's life, with answer options of "not at all," "a little," "somewhat," "quite a bit," and "very much." The final question asks "if you were to spend the rest of your life with your dry mouth/throat dryness just the way it is now, how would you feel about this?" and includes options ranging from "delighted" to "terrible." All 15 questions can be translated to a score of 0-4, with a score of 4 indicating the most dry mouth-related problems and 0 indicating no dry mouth-related problems.
Quality of life as assessed by the Xerostomia Quality of Life Scale (XeQoLS) | 30 months after baseline visit
  The XeQoLS consists of 15 questions. The first 14 questions assess how dryness in the mouth impacts the individual's life, with answer options of "not at all," "a little," "somewhat," "quite a bit," and "very much." The final question asks "if you were to spend the rest of your life with your dry mouth/throat dryness just the way it is now, how would you feel about this?" and includes options ranging from "delighted" to "terrible." All 15 questions can be translated to a score of 0-4, with a score of 4 indicating the most dry mouth-related problems and 0 indicating no dry mouth-related problems.
Quality of life as assessed by the Oral Health Related Quality of Life (OHRQoL) | Baseline
  Oral health related quality of life will be assessed using the questionnaire developed for the National Health and Nutrition Examination Survey (NHANES). This questionnaire assesses the topic areas of last visit to dentist or lack of dental care; direct conversation with dental professional about your dental health; dental health perception; oral cancer exam; use of dental floss or dental rinse product; and periodontal disease self-report. Each topic area uses a separate scoring system and may be assessed individually.
Quality of life as assessed by the Oral Health Related Quality of Life (OHRQoL) | 12 months after baseline visit
  Oral health related quality of life will be assessed using the questionnaire developed for the National Health and Nutrition Examination Survey (NHANES). This questionnaire assesses the topic areas of last visit to dentist or lack of dental care; direct conversation with dental professional about your dental health; dental health perception; oral cancer exam; use of dental floss or dental rinse product; and periodontal disease self-report. Each topic area uses a separate scoring system and may be assessed individually.
Quality of life as assessed by the Oral Health Related Quality of Life (OHRQoL) | 24 months after baseline visit
  Oral health related quality of life will be assessed using the questionnaire developed for the National Health and Nutrition Examination Survey (NHANES). This questionnaire assesses the topic areas of last visit to dentist or lack of dental care; direct conversation with dental professional about your dental health; dental health perception; oral cancer exam; use of dental floss or dental rinse product; and periodontal disease self-report. Each topic area uses a separate scoring system and may be assessed individually.
Quality of life as assessed by the Oral Health Related Quality of Life (OHRQoL) | 30 months after baseline visit
  Oral health related quality of life will be assessed using the questionnaire developed for the National Health and Nutrition Examination Survey (NHANES). This questionnaire assesses the topic areas of last visit to dentist or lack of dental care; direct conversation with dental professional about your dental health; dental health perception; oral cancer exam; use of dental floss or dental rinse product; and periodontal disease self-report. Each topic area uses a separate scoring system and may be assessed individually.
Quality of life as assessed by the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool | Baseline
  The TAPS tool screens for substance use (including tobacco, alcohol, prescription medication, and other drugs) and includes a brief assessment of abuse risk for those who screen positive. Individuals who screen positive for use of any of the substances are then scored as 0 (no use in the past 3 months), 1 (problem use), and 2+ (high risk for substance use disorder).
Quality of life as assessed by the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool | 12 months after baseline visit
  The TAPS tool screens for substance use (including tobacco, alcohol, prescription medication, and other drugs) and includes a brief assessment of abuse risk for those who screen positive. Individuals who screen positive for use of any of the substances are then scored as 0 (no use in the past 3 months), 1 (problem use), and 2+ (high risk for substance use disorder).
Quality of life as assessed by the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool | 24 months after baseline visit
  The TAPS tool screens for substance use (including tobacco, alcohol, prescription medication, and other drugs) and includes a brief assessment of abuse risk for those who screen positive. Individuals who screen positive for use of any of the substances are then scored as 0 (no use in the past 3 months), 1 (problem use), and 2+ (high risk for substance use disorder).
Quality of life as assessed by the Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS) Tool | 30 months after baseline visit
  The TAPS tool screens for substance use (including tobacco, alcohol, prescription medication, and other drugs) and includes a brief assessment of abuse risk for those who screen positive. Individuals who screen positive for use of any of the substances are then scored as 0 (no use in the past 3 months), 1 (problem use), and 2+ (high risk for substance use disorder).

SECONDARY OUTCOMES:
Xerostomia as assessed by stimulated saliva secretion rate | Baseline
  Prevalence of xerostomia
Xerostomia as assessed by stimulated saliva secretion rate | 6 months after baseline visit
  Prevalence of xerostomia
Xerostomia as assessed by stimulated saliva secretion rate | 12 months after baseline visit
  Prevalence of xerostomia
Xerostomia as assessed by stimulated saliva secretion rate | 18 months after baseline visit
  Prevalence of xerostomia
Xerostomia as assessed by stimulated saliva secretion rate | 24 months after baseline visit
  Prevalence of xerostomia
Xerostomia as assessed by stimulated saliva secretion rate | 30 months after baseline visit
  Prevalence of xerostomia
Saliva proteins | Baseline
  levels of amylase expression will be assessed
Saliva proteins | 6 months after baseline visit
  levels of amylase expression will be assessed
Saliva proteins | 12 months after baseline visit
  levels of amylase expression will be assessed
Saliva proteins | 18 months after baseline visit
  levels of amylase expression will be assessed
Saliva proteins | 24 months after baseline visit
  levels of amylase expression will be assessed
Saliva proteins | 30 months after baseline visit
  levels of amylase expression will be assessed
Saliva proteins | baseline visit
  levels of IgA expression will be assessed
Saliva proteins | 6 months after baseline visit
  levels of IgA expression will be assessed
Saliva proteins | 12 months after baseline visit
  levels of IgA expression will be assessed
Saliva proteins | 18 months after baseline visit
  levels of IgA expression will be assessed
Saliva proteins | 24 months after baseline visit
  levels of IgA expression will be assessed
Saliva proteins | 30 months after baseline visit
  levels of IgA expression will be assessed
Correlative measures | Baseline through 30 months
  Salivary cytokines: levels of IL-6, IL-7, IL-10, TNF-α, neopterin, β-2-microglobulin (β2M) and monocyte chemotactic protein-1 will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Temitope Omolehinwa, BDS, DScD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omolehinwa TT, Akintoye SO, Gabinskiy M, Lo Re V 3rd, Mupparapu M, Urbina R, Schaubel DE, Corby PM. Oral health outcomes in an HIV cohort with comorbidities- implementation roadmap for a longitudinal prospective observational study. BMC Oral Health. 2023 Oct 17;23(1):763. doi: 10.1186/s12903-023-03527-5. PMID 37848867